CLINICAL TRIAL: NCT06681077
Title: I Can Join the Fight Against Cancer: An Intervention to Programmatically Build Grassroots Actions to Reduce the Cancer Burden
Brief Title: A Community Health Education Intervention for Increasing Community-driven Actions to Reduce the Cancer Burden in Western New York
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 4186824; NCI-2024-09012 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 4186824 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (I CAN intervention) (Experimental): Participants attend an I CAN intervention workshop over 2 hours.
  Interventions: Procedure: Community Health Education; Other: Survey Administration

INTERVENTIONS:
Procedure: Community Health Education — Receive I CAN intervention
  Other Names: Community Education
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates a community health education intervention (I CAN) for increasing community-driven actions to reduce the cancer burden in Western New York. Engaging community members is a critical component of designing impactful programs to reduce the cancer burden. Leaders at the national, state, and local levels have all called for more community partnerships and engagement in design of health intervention and policies. The I CAN intervention is a workshop that includes a presentation outlining key concepts related to social network processes and the cancer burden in Western New York, a structured skill-building activity, and then empowering and motivating activities meant to cultivate momentum and excitement for action. This community health education intervention may be able to provide a formalized process for empowering and facilitating community members to take steps to reduce the community cancer burden.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the feasibility of the I CAN intervention. II. Examine the acceptability of the I CAN intervention. III. Examine topic areas selected for action within participants' I CAN plans for action.

OUTLINE:

Participants attend an I CAN intervention workshop over 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Able to participate in English

Exclusion Criteria:

* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Demand | Up to 2 years
  Feasibility will be assessed through demand, which will be evaluated as the number of people enrolled and the demographics of participants. Descriptive analyses will be used.
Practicality | Up to 2 years
  Practicality will be assessed through the percentage of participants who complete different aspects of the intervention. Descriptive analyses will be used.
Acceptability | UP to 2 years
  Acceptability will be examined through post-intervention measures, including the Acceptability of Intervention Measure, Intervention Appropriateness Measure, and Feasibility of Intervention Measure. Descriptive analyses will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bouchard, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States